CLINICAL TRIAL: NCT07304674
Title: The Association Between Primary Aldosteronism and Cognitive Dysfunction
Acronym: PACD
Status: Recruiting | Type: Observational
Sponsor: Xinjiang Medical University (Other)
Responsible Party: Principal Investigator, Xiang Xie, Professor, Xinjiang Medical University
Other Study IDs: K202511-02
Record Dates: First submitted 2025-12-13; First posted 2025-12-26 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2026-01

CONDITIONS: Primary Aldosteronism; Cognitive Dysfunction; Mild Cognitive Impairment (MCI); Dementia
MeSH Terms: conditions — Hyperaldosteronism; Cognitive Dysfunction; Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn about the prevalence, progression, and influencing factors of cognitive impairment in patients with primary aldosteronism (PA). The main questions it aims to answer are:

1. What is the prevalence of baseline cognitive impairment in PA patients and what factors are associated with it?
2. What is the incidence of cognitive progression in PA patients within 1 and 5 years of follow-up and what factors influence this progression? Participants who are already diagnosed with PA as part of their regular medical care will be invited to join this long-term study. They will complete regular cognitive tests, medical check-ups, and questionnaires for up to 5 years. Some participants will also have optional blood tests and brain scans to help researchers understand the causes behind any cognitive changes.

DETAILED DESCRIPTION:
This is a prospective observational cohort study conducted in two tertiary hospitals. The main purposes are to investigate the prevalence and influencing factors of mild cognitive impairment (MCI) and dementia at baseline in patients with primary aldosteronism (PA), assess the incidence and influencing factors of cognitive progression within 1 and 5 years of follow-up, and compare exploratory biomarkers, such as plasma neurofilament light chain (NfL) and brain magnetic resonance imaging (MRI) measures, between PA patients with and without baseline cognitive impairment. Eligible patients will be followed up for 5 years, with regular cognitive function assessment, clinical indicator monitoring, and detection of relevant biomarkers and imaging indicators. The study aims to delineate the cognitive trajectory in PA and identify associated clinical and biological predictors.

ELIGIBILITY:
Inclusion Criteria:

* 1. Aged ≥ 40 years.
* 2. Biochemically confirmed diagnosis of Primary Aldosteronism (PA) according to contemporary guidelines (e.g., confirmed positive case detection test and confirmatory test).
* 3. Ability to understand and cooperate with comprehensive neuropsychological assessment.
* 4. Voluntary participation and provision of written informed consent.

Exclusion Criteria:

* 1. Significant visual, hearing, or motor impairment that prevents completion of cognitive testing.
* 2. History of major neurological disorders (e.g., stroke, Parkinson's disease, intracranial tumor, severe traumatic brain injury).
* 3. History of major psychiatric illness, intellectual disability, or current use of antipsychotic medications.
* 4. Diagnosis of secondary hypertension other than PA.
* 5. Unwillingness to participate by the patient or their legal representative.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will establish a prospective, two-center cohort of primary aldosteronism (PA). Designed to capture the full baseline spectrum of cognitive function, the cohort aims to systematically determine the incidence and progression of cognitive impairment and identify its clinical and biochemical predictors.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-12-31 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
1-Year Early Cognitive Progression in Patients with PA | Baseline and 12 months.
  Defined as the proportion of PA patients who experience cognitive progression within 1 year of follow-up. Cognitive progression includes three transitions: 1) Normal cognition → MCI; 2) Normal cognition → Dementia; 3) MCI → Dementia.The diagnostic criteria for MCI and dementia are based on the National Institute on Aging-Alzheimer's Association (NIA-AA) criteria (for MCI and dementia). All events are adjudicated by an independent endpoint committee.
5-Year Cumulative Incidence of Cognitive Progression in Patients with PA | Baseline, 12, 24, 36, 48, and 60 months.
  Defined as the proportion of PA patients who experience cognitive progression within 5 years of follow-up. Cognitive progression follows the same transitions and diagnostic criteria as the 1-year primary outcome (NIA-AA criteria). All events are adjudicated by an independent endpoint committee.

SECONDARY OUTCOMES:
Baseline Prevalence of Cognitive Impairment (MCI or Dementia) in Patients with PA | Baseline
  The proportion of patients with PA who have MCI or dementia at study baseline, as adjudicated by an independent endpoint committee using the NIA-AA criteria.
3-year cumulative incidence of cognitive progression in patients with PA | Baseline, 12, 24, and 36 months.
  The proportion of patients who experience cognitive progression within 3 years of follow-up. Cognitive progression is defined as the same transitions and diagnostic criteria (NIA-AA) as the primary outcomes.
Longitudinal Change in Global Cognitive Function | Baseline, 12, 24, 36, 48, and 60 months
  Change in global cognitive function as measured by the validated Chinese version of the Montreal Cognitive Assessment (MoCA, Beijing version). The total score ranges from 0 to 30 (higher scores indicate better cognitive function).
Change in Functional Activities Questionnaire (FAQ) total score | Baseline, 12, 24, 36, 48, and 60 months.
  Change in the total score of the validated Chinese version of the FAQ (range 0-30; higher scores indicate greater impairment). This scale assesses instrumental activities of daily living.
Change in Neuropsychiatric Inventory (NPI) Total Score | Baseline, 12, 24, 36, 48, and 60 months.
  Change in the validated Chinese version of the NPI total score (range: 0-144; higher scores indicate greater neuropsychiatric symptom burden), assessing 12 behavioral domains.
Office Blood Pressure Control Rate | 12, 24, 36, 48, and 60 months.
  The proportion of patients achieving controlled office blood pressure at each post-baseline follow-up visit. Control is defined as an average of triplicate seated measurements with systolic blood pressure (SBP) < 140 mmHg and diastolic blood pressure (DBP) < 90 mmHg.
24-Hour Ambulatory Blood Pressure Control Rate | 12, 24, 36, 48, and 60 months.
  The proportion of patients achieving controlled 24-hour ambulatory blood pressure. Control is defined as a mean 24-hour SBP < 130 mmHg and DBP < 80 mmHg.
Plasma Aldosterone Concentration (PAC) | Baseline, 12, 24, 36, 48, and 60 months.
  Absolute plasma aldosterone concentration, measured in pg/mL.
Plasma Renin Concentration (PRC) | Baseline, 12, 24, 36, 48, and 60 months.
  The absolute concentration of renin in plasma, measured in pg/mL. This outcome, along with aldosterone, is used to calculate the aldosterone-to-renin ratio (ARR), a key screening and diagnostic biomarker for PA.
Serum Potassium (K+) Level | Baseline, 12, 24, 36, 48, and 60 months.
  Absolute serum potassium concentration, measured in mmol/L.
Serum Sodium (Na+) Level | Baseline, 12, 24, 36, 48, and 60 months.
  Absolute serum sodium concentration, measured in mmol/L.
Low-Density Lipoprotein Cholesterol (LDL-C) Level | Baseline, 12, 24, 36, 48, and 60 months.
  Fasting serum concentration of LDL-C, measured in mmol/L.
Lipoprotein(a) (Lp(a)) Level | Baseline, 12, 24, 36, 48, and 60 months.
  Fasting serum concentration of Lp(a), measured in nmol/L, an independent risk factor for cardiovascular disease.
Fasting Plasma Glucose Level | Baseline, 12, 24, 36, 48, and 60 months.
  Concentration of glucose in plasma after ≥8 hours of fasting, measured in mmol/L.
Glycated Hemoglobin (HbA1c) Level | Baseline, 12, 24, 36, 48, and 60 months.
  The percentage of HbA1c in blood, reflecting average blood glucose over the preceding 2-3 months.
Estimated Glomerular Filtration Rate (eGFR) | Baseline, 12, 24, 36, 48, and 60 months.
  Renal function assessed by the eGFR, calculated from serum creatinine using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation (units: mL/min/1.73m²).
Urinary Albumin-to-Creatinine Ratio (UACR) | Baseline, 12, 24, 36, 48, and 60 months.
  The UACR measured from a spot urine sample and reported in mg/g, a marker of kidney damage.
Left Ventricular Mass Index (LVMI) | Baseline, 12, 24, 36, 48, and 60 months.
  Left ventricular mass indexed to body surface area (g/m²), calculated from echocardiographic measurements. The key criterion for diagnosing left ventricular hypertrophy.
Left Ventricular Ejection Fraction (LVEF) | Baseline, 12, 24, 36, 48, and 60 months.
  The percentage of blood ejected from the left ventricle during each contraction, measured by echocardiography.
Carotid Intima-Media Thickness (CIMT) | Baseline, 12, 24, 36, 48, and 60 months.
  The mean far-wall intima-media thickness of the common carotid artery (mm), measured bilaterally by ultrasound. A marker of subclinical atherosclerosis.
Plasma NfL Concentration (Sub-study) | Baseline, 12, 36, and 60 months.
  Concentration of plasma NfL (pg/mL), a biomarker of neuroaxonal injury, measured in a pre-defined sub-cohort.
White Matter Hyperintensity (WMH) Volume (Sub-study) | Baseline, 12, 36, and 60 months.
  Total volume of white matter hyperintensities, quantified in cubic millimeters (mm³) from T2-fluid-attenuated inversion recovery (FLAIR) magnetic resonance imaging sequences. WMH volume is a quantitative marker of cerebral small vessel disease burden.
Cerebral Blood Flow (Sub-study) | Baseline, 12, 36, and 60 months.
  Quantitative measurement of regional and global cerebral blood flow, obtained via arterial spin labeling (ASL) magnetic resonance imaging, and reported in milliliters per 100 grams of tissue per minute (mL/100g/min).
Incidence of Major Adverse Cardiovascular Events (MACE) | Baseline, 12, 24, 36, 48, and 60 months.
  The proportion of patients who experience an adjudicated MACE, a composite of non-fatal myocardial infarction, non-fatal stroke, hospitalization for heart failure, or cardiovascular death.
All-cause mortality | Baseline, 12, 24, 36, 48, and 60 months.
  Record of deaths from any cause during follow-up. Confirmed by medical records, family follow-up, or national death registration systems.

CONTACTS AND LOCATIONS:
Overall Officials: Xiang Xie, PhD, Study Chair — First Affiliated Hospital of Xinjiang Medical University
Locations (2):
- China (2):
  - The First Affiliated Hospital of Chengdu Medical College, Chengdu, Sichuan
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang

IPD SHARING:
Plan to Share IPD: No